CLINICAL TRIAL: NCT04139161
Title: Cycling Intervention on Symptoms of Patients With Knee Osteoarthritis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: The University of Tennessee, Knoxville (Other)
Responsible Party: Principal Investigator, Tanner Thorsen, Graduate Research Assistant, The University of Tennessee, Knoxville
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UTK IRB-19-05254-XP
Record Dates: First submitted 2019-10-22; First posted 2019-10-25 (Actual); Last update posted 2020-04-07 (Actual); Status verified 2020-04

CONDITIONS: Osteoarthritis, Knee
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Q-Factor Intervention (Experimental): Participants will progress through three increasing Q-Factors for each cycling workrate; Q-Factor 1 (Q1, 192mm), Q2 (234mm), Q3 (276mm). After completing bouts of all three Q-Factors for a given workrate, workrate will be increased by 20 Watts and bouts at each Q-Factor will be repeated.
  Interventions: Procedure: Q-Factor Intervention

INTERVENTIONS:
Procedure: Q-Factor Intervention — The intervention period will consist of 12 training sessions across four consecutive weeks, with three training sessions held per week. If pain is not increased or reduced and Rating of Perceived Exertion is ≤12, the participant will progress to the next bout. If pain is increased from the pre-bout pain score, participants will repeat the bout, at the same workrate and Q-Factor settings. Following this fashion, participants will progress through three increasing Q-Factors for each given workrate; Q-Factor 1 (Q1, 192mm), Q2 (234mm), Q3 (276mm). After completing bouts of all three Q-Factors for a given workrate, workrate will be increased by 20 Watts and bouts at each Q-Factor will be repeated. For each training session, participants will complete bouts of cycling until 1) the maximum number of bouts (4 bouts) has been accomplished, 2) self-reported Rating of Perceived Exertion >12, indicating a transition to moderate physical activity, or 3) self-reported pain >5.

SUMMARY:
This study is designed to determine the effect of a cycling training program which modulates frontal and sagittal plane knee joint loading with graded increases of Q-Factor and cycling workrate in persons with symptomatic knee osteoarthritis.

DETAILED DESCRIPTION:
The knee joint is one of the most common joints affected by osteoarthritis, and knee osteoarthritis is primarily observed in the medial compartment. This is in part attributable to the increased load experienced by the medial compartment during level walking. Patients with symptomatic knee osteoarthritis exhibit altered gait mechanics; namely a reduced loading response knee extension moment and an increased internal knee abduction moment. As a surrogate measure for medial compartment joint loading, loading response knee abduction moment in level walking has been shown to increase with the severity of knee osteoarthritis.

Recent gait modification research has shown that increased step-width decreases peak Knee abduction moment for persons with knee osteoarthritis. The inter-pedal width of a bicycle or cycle ergometer, known as Q-Factor, is analogous in cycling to step-width in gait. In contrast to gait, increased Q-Factor has been shown to increase the knee abduction moment during stationary cycling. Modulating sagittal and frontal plane loading of the knee in a graded manner during cycling may promote healthy adaptation to muscle weakness and pain. This adaptation may be manifest through restoration of altered knee joint biomechanics (knee extension moment, knee abduction moment), which, in turn, may also provide benefit to gait mechanics.

ELIGIBILITY:
Inclusion Criteria:

* Men and Women between the ages of 50 and 75 years old.
* Diagnosed with medial compartment tibiofemoral osteoarthritis in one of their knees.
* Be able to walk unaided for at least 25 consecutive minutes.
* Present with knee pain for at least 6 months occurring on a majority of the days in the month, or on most days (more than or equal to 4 of 7 days in a week) in one or both knees for at least 4 months.
* Osteophytes on knee x-rays.
* Grade 2 or higher out of a maximum of 4 on a modified Kellgren/Lawrence grade on the knee radiograph.

Exclusion Criteria:

* Initial Visual Analog Scale pain scores greater than 7.
* Diagnosed osteoarthritis of ankles, hips, or symptomatic osteoarthritis of the spine.
* Arthroplasty of any other lower extremity joint.
* BMI value greater than 40 kg/m2.
* Any major lower extremity injury in the past 6 months.
* Systemic Inflammatory Arthritis.
* Systemic Pain Conditions.
* Neurological Conditions that impact gait or cycling.
* Pregnant or Nursing Women.
* Major cardiovascular disease with an exercise limitation prescribed by a physician.
* Steroid injection at the knee within the previous 3 months.

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2019-12-17 (Actual); Primary Completion 2021-05-31 (Estimated); Study Completion 2021-05-31 (Estimated)

PRIMARY OUTCOMES:
Knee Abduction Moment - Cycling | Baseline, 1 month, 2 month
  Change in Knee Extension Moment during cycling.
Knee Abduction Moment - Gait | Baseline, 1 month, 2 month
  Change in Knee Extension Moment during gait.

SECONDARY OUTCOMES:
Visual Analog Pain | Immediately following exercise (walking and cycling).
  Self-Reported pain intensity during gait and cycling reported on a scale from 1-10 with higher scores reflecting more pain.
Knee Extension Moment - Cycling | Baseline, 1 month, 2 month
  Change in Knee Extension Moment during cycling
Knee Extension Moment - Gait | Baseline, 1 month, 2 month
  Change in Knee Extension Moment during Gait
Knee Injury and Osteoarthritis Outcome Score | Baseline, 1 month, 2 month
  Change in Knee Injury and Osteoarthritis Outcome Score reported on a scale from 0 to 100, with 0 representing extreme problems and 100 representing no problems.

CONTACTS AND LOCATIONS:
Overall Officials: Tanner Thorsen, MS, Principal Investigator — University of Tennessee, Knoxville
Locations (1):
- Biomechanics/Sports Medicine Lab, Knoxville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No